CLINICAL TRIAL: NCT02671682
Title: Immunoadsorption vs. Plasmapheresis in the Escalation Therapy of Relapse in Multiple Sclerosis and Clinically Isolated Syndrome
Brief Title: Immunoadsorption vs. Plasmapheresis in the Escalation Therapy of Relapse in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Christian Ludolph, Prof. (Other)
Responsible Party: Sponsor-Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAPEMS
Record Dates: First submitted 2016-01-22; First posted 2016-02-02 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Immunoadsorption; Plasmapheresis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunoadsorption (Experimental): Immunoadsorption on 5 consecutive days with protein A columns and 2,5-fold patient's plasma volume
  Interventions: Procedure: Immunoadsorption
- Plasmapheresis (Active Comparator): Plasmapheresis on 5 consecutive days with 2l plasma exchange
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Procedure: Immunoadsorption
  Arms: Immunoadsorption
Procedure: Plasmapheresis
  Arms: Plasmapheresis

SUMMARY:
This observational study investigates the efficacy and safety of immunoadsorption versus plasmapheresis in 60 patients with relapse in Multiple Sclerosis and Clinically isolated syndrome who do not fully recover after a high doses of intravenous corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* relapse of Multiple Sclerosis or Clinically Isolated Syndrome (without complete remission after high dose steroid therapy)
* informed consent
* age ≥ 12 years old

Exclusion Criteria:

* clinical or laboratory signs of infection
* intake of Angiotensin Converting Enzyme Inhibitor within 1 week prior to first treatment

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) | 4 weeks

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 2 and 4 weeks
EuroQol (EQ5D-5L) | 2 and 4 weeks
Response Rate | 4 weeks
  defined as share of patients who show an improvement of least 10% in MSFC (see Outcome 1) compared to baseline value
Vision | 4 weeks
  defined as percentage of normal vision as measured by visual test according to EDSS standardized testing (see outcome 2)
Visually Evoked Potentials (VEP; P100 latency) | 4 weeks
Somatosensory Evoked Potentials (SEP; Medianus and Tibialis; N20-, P40-latency) | 4 weeks
Thickness of Retinal Nerve Fiber Layer (RNFL) in Optical Coherence Tomography (OCT) | 4 weeks
Verbaler Lern- und Merkfähigkeitstest (VLMT) score | 4 weeks
MSFC | 2 weeks
Thickness of Ganglion Cell Layer (GCL) in OCT | 4 weeks
Symbol Digit Modalities Test (SDMT) score | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vardakas I, Dorst J, Huss A, Mayer B, Fangerau T, Taranu D, Tumani H, Senel M. Serum neurofilament light chain and glial fibrillary acidic protein for predicting response to apheresis in steroid-refractory multiple sclerosis relapses. Eur J Neurol. 2024 Aug;31(8):e16323. doi: 10.1111/ene.16323. Epub 2024 May 3. PMID 38700322
- [Derived] Dorst J, Fangerau T, Taranu D, Eichele P, Dreyhaupt J, Michels S, Schuster J, Ludolph AC, Senel M, Tumani H. Safety and efficacy of immunoadsorption versus plasma exchange in steroid-refractory relapse of multiple sclerosis and clinically isolated syndrome: A randomised, parallel-group, controlled trial. EClinicalMedicine. 2019 Nov 14;16:98-106. doi: 10.1016/j.eclinm.2019.10.017. eCollection 2019 Nov. PMID 31832624